CLINICAL TRIAL: NCT03621111
Title: Adherence, Pharmacists and Secondary Prevention in Acute Myocardial Infarction: A Pilot Controlled Clinical Trial on the Role of Community Pharmacist in Monitoring Medication Adherence and Improving Clinical Outcomes in Post-infarction
Brief Title: A Trial on the Role of Community Pharmacist in Improving Adherence and Clinical Outcomes in Post-Infarction
Acronym: IM-ADHERENCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda ULSS 5 Polesana (Other)
Collaborators: University of Padova (Other)
Responsible Party: Principal Investigator, Raffaella Ruzza, Hospital Pharmacist, Azienda ULSS 5 Polesana
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017/18
Record Dates: First submitted 2018-07-18; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Myocardial Infarction, Acute; ST Segment Elevation Myocardial Infarction; Non-ST Elevation Myocardial Infarction (nSTEMI)
Keywords: Myocardial Infarct; Medication Adherence; Community Pharmacist; Patient counseling; Pill counts; Hospital re-admission; Antiplatelet therapy; Beta-blockers; Lipid-lowering therapy; Angiotensin-Converting Enzyme Inhibitors (ACEi); Renin Angiotensin System Inhibitors (RASi); Mineralocorticoid/aldosterone receptor antagonists
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adherence plan (Experimental): At the discharge, the hospital pharmacist will complete the medication reconciliation and assess the patient's medications. All patients enrolled will undergo three interventions in order to improve medication adherence: counseling, pill counts and self-questionnaire. The adherence plan concerns 6 classes of drugs recommended by the European Society of Cardiology in acute myocardial infarction. The adherence plan is performed by the community pharmacists. The hospital pharmacist will complete the discharge care form for the community pharmacist who has in charge the patient. Each patient will be scheduled for the first meeting with his community pharmacist within one month from the hospital discharge; afterward the adherence plan will be submitted every 3 months.
  Interventions: Behavioral: Patient-counseling; Behavioral: Patient self-administered questionnaire; Behavioral: Pills counts
- Control group (No Intervention): All the patients discharged from the cardiological ward between September 2017 and February 2018 with a primary diagnosis of acute myocardial infarction has been enrolled in the control arm. These patients have been discharged with the current standard therapy and without any adherence plan performed by the community pharmacists. The investigators will collect the data from the administrative pharmaceutical databases throughout 12 months from the hospital discharge.

INTERVENTIONS:
Behavioral: Patient-counseling — After one month from the hospital discharge, the pharmacist will give to the patient general advices and suggestions regarding disease, therapy and drugs.
  Arms: Adherence plan
Behavioral: Patient self-administered questionnaire — The pharmacist will submit the questionnaire to the patient for the evaluation of drug adherence, life style, feelings and approach to therapies, at 30 days, 3, 6, 9 and 12 months from the enrollment. This self-questionnaire of 13 questions contains the 8 multiple choice questions of the Morisky medication adherence scale (MMAS-8-Item, Italian version).
  Arms: Adherence plan
Behavioral: Pills counts — At the time of the monthly drug re-supply at the community pharmacy, the patient will bring the boxes of the drugs taken in the previous month (empty or not), for the pill counts. The pharmacist will verify the correct assumption of the pharmacological therapies.
  Arms: Adherence plan

SUMMARY:
The purpose of this pilot study is to evaluate the effectiveness of the active involvement of Community Pharmacists in improving adherence to medical prescriptions in patients with acute myocardial infarction (AMI), reducing the rate of adverse events and / or re-admissions due to cardiovascular disease and reducing overall health costs. The Hospital and Community Pharmacists will collaborate with each other, the patients, heart specialists and primary care physicians, throughout 12 months from the hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Discharged with a primary diagnosis of Acute Myocardial Infarction (AMI, ICD-9 code: 410.x1) from a cardiological ward;
* Required treatment with antiplatelet therapy, beta-blockers, lipid-lowering therapy, Angiotensin-Converting Enzyme Inhibitors (ACEi), Renin Angiotensin System Inhibitors (RASi) and/or mineralocorticoid/aldosterone receptor antagonists at the hospital admission, alone or in combination;
* Agreeable to participate in adherence plan (if randomized to interventional arm) performed by the community pharmacist who has in charge the patient;
* Agreeable to understand and accept the purpose of the study;
* Signed of the informed consent to participate;
* Be complying with the protocols' procedures within the entire period of study.

Exclusion Criteria:

* Any prior history of acute myocardial infarction within 6 months prior to study entry;
* Presence of physical or cognitive impairment or dementia;
* Permanent long-term residence in Hospice or facility residents;
* History or presence of any other cardiovascular disease with a life expectancy of < 1 year, hypertension excluded.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-02-19 (Estimated); Study Completion 2019-08-19 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in medication adherence after 6 months in the interventional and control arms | baseline, 6 months
  Change in medication adherence as measured by the calculation of Proportion of Days Covered (PDC) in the two arms. The value of PDC will be compared with the results of the pill counts performed by the community pharmacist. The endpoint concerns all medications recommended by the European Society of Cardiology for the treatment of AMI. The composite PDC will be an average of the individual PDC for each drug class

SECONDARY OUTCOMES:
Change from baseline in medication adherence after 12 months in the interventional and control arms | baseline, 12 months
  Change in medication adherence as measured by the calculation of Proportion of Days Covered (PDC) in the two arms
Change in re-admission rates due to cardiovascular events after 12 months between the interventional arm and the control arm | 12 months
  Rates of hospital re-admission in the two arms: any re-admission identified by the heart specialist and due to cardiovascular events will be categorized based on the International Classification of Diseases (ICD)-9 classification. The rate will be measured as the per cent ratio of the re-admissions in the interventional arm and the re-admissions in the control arm

OTHER OUTCOMES:
Change in health care costs over 12 months in the interventional and control arms | 12 months
  Change in average (mean) health care costs as measured by calculation of hospitalization and medication costs over 12 months for each patient in the interventional and control arms. The hospitalization and medication costs are assessed by the administrative pharmaceutical databases
Change from baseline in adherence scores on the Morisky medication adherence scale after 12 months in the interventional arm | baseline, 12 months
  Change in medication adherence as assessed by the Morisky medication adherence scale (MMAS) in the interventional arm. The MMAS is an international validated scale to assess the patient's medication adherence in chronic diseases. Each patient will answer the 8 multiple choice questions of the MMAS by completing the self-questionnaire every 3 months
Prescriptions of fixed dose drug combinations in the interventional and control arms | baseline, 12 months
  Number of patients with one or more prescriptions of fixed dose drug combinations (FDCs) as measured by total months' supply dispensed in the interventional and control arms
Description of pluri-pharmacological therapies in the interventional and control arms | 12 months
  Change from baseline in drugs' prescriptions as assessed by the administrative pharmaceutical databases. This is calculated by analysing drugs' prescriptions for both myocardial infarction and other chronic co-morbidities (such as hypertension, diabetes)

CONTACTS AND LOCATIONS:
Overall Officials: Raffaella Ruzza, University, Principal Investigator — Azienda ULSS 5 Polesana; Erika Vighesso, University, Principal Investigator — University of Padova; Gianni Bregola, University, Principal Investigator — Azienda ULSS 5 Polesana
Locations (1):
- Azienda ULSS 5 Polesana, Rovigo, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Investigators are committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent Ethics Committee on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.

REFERENCES:
- [Background] Gujral G, Winckel K, Nissen LM, Cottrell WN. Impact of community pharmacist intervention discussing patients' beliefs to improve medication adherence. Int J Clin Pharm. 2014 Oct;36(5):1048-58. doi: 10.1007/s11096-014-9993-y. Epub 2014 Aug 19. PMID 25135805
- [Result] Roffi M, Patrono C, Collet JP, Mueller C, Valgimigli M, Andreotti F, Bax JJ, Borger MA, Brotons C, Chew DP, Gencer B, Hasenfuss G, Kjeldsen K, Lancellotti P, Landmesser U, Mehilli J, Mukherjee D, Storey RF, Windecker S; ESC Scientific Document Group. 2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: Task Force for the Management of Acute Coronary Syndromes in Patients Presenting without Persistent ST-Segment Elevation of the European Society of Cardiology (ESC). Eur Heart J. 2016 Jan 14;37(3):267-315. doi: 10.1093/eurheartj/ehv320. Epub 2015 Aug 29. No abstract available. PMID 26320110
- [Result] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Result] Ho PM, Spertus JA, Masoudi FA, Reid KJ, Peterson ED, Magid DJ, Krumholz HM, Rumsfeld JS. Impact of medication therapy discontinuation on mortality after myocardial infarction. Arch Intern Med. 2006 Sep 25;166(17):1842-7. doi: 10.1001/archinte.166.17.1842. PMID 17000940
- [Result] Ryan R, Santesso N, Lowe D, Hill S, Grimshaw J, Prictor M, Kaufman C, Cowie G, Taylor M. Interventions to improve safe and effective medicines use by consumers: an overview of systematic reviews. Cochrane Database Syst Rev. 2014 Apr 29;2014(4):CD007768. doi: 10.1002/14651858.CD007768.pub3. PMID 24777444